CLINICAL TRIAL: NCT05787808
Title: The Effect on Bone Marker and Body Mineral Density (BMD) of Daily Jarlsberg Cheese Intake in Risk Patient for Osteoporosis
Brief Title: Profylactic Treatment for Patients in Risk Osteoporosis
Acronym: PF-Jarlsberg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Collaborators: Tine (Industry); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor Emeritus, Meddoc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PF-Jarlsberg/IIIA; 2022-003252-13 (EudraCT Number)
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Osteopenia or Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: The patients are randomised (1:1) into to parallel groups and followed up in 16 weeks. All the patients are switched to the same treatment for the following 16 weeks
Masking Description: Masking is not posible in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Active Comparator): 1000 mg Calcium tablets + 20µg vitamin D and optimal efficacy dose of Jarlsberg cheese
  Interventions: Dietary Supplement: Calsium, Vitamin D, Jarlsberg cheese
- Treatment 2 (Active Comparator): 1000 mg Calcium tablets + 20µg vitamin D
  Interventions: Dietary Supplement: Calsium, Vitamin D, Jarlsberg cheese

INTERVENTIONS:
Dietary Supplement: Calsium, Vitamin D, Jarlsberg cheese — Oral

SUMMARY:
The aim is to compare the daily intake of Calsium (Ca) + vitamin D with and without daily optimal efficacy dose (OED) of Jarlsberg on Bone Mineral Density (BMD) and bone markers (BM) to Osteopeni patients (OP).

* The study population consists of OP-patients of post-menopausal women and men above 55 years of age. OP patients are defined as patients with a T-score below 0.0, but larger than -2.5.
* The study will be performed as a randomized, single-blinded Norwegian multicentre trial with stratified semi-cross-over design with gender and site as stratification factors. The OP-patients included in the study will be allocated to one of the two treatment groups by block randomization with random block size between 2 and 6.
* Women in post-menopausal age have a daily OED Jarlsberg of 45 gram and men in the same age interval have a daily OED of 55 gram.
* The main response variable will be the change in Bone Mineral Density (BMD),total Osteocalcin (tOC) and different bone markers (BM).
* Participants, who fulfil the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will be included and receiving 40µg vitamin D and 500 mg Ca tablets per day, but asked not to eat Jarlsberg cheese the following week. During this week demographic data, bloodsampling for measurement of Osteocalcin and BM and diet registration will be performed.In the clinical study, all the included patients will continue with Ca+ vitamin D, but half of the patient will additionally receive daily OED of Jarlsberg cheese. After 16 weeks, all the patients will receive both Ca+vitamin D and OED of Jarlsberg for addionally 16 weeks. The total duration of the study will be 32 weeks for the patients initially allocated to Jarlsberg and 48 weeks for those allocated only to Ca+vitamin D. The patients will be investigated initially and every 16 weeks.
* A total of 30 patients will be included in each of the two groups.

DETAILED DESCRIPTION:
Aim

* To estimate the effect of daily optimal efficacy dose (OED) of Jarlsberg cheese on BMD and bone markers to patients with Osteopeni (OP).
* To compare daily intake of Calsium (Ca) and vitamin D with and without OED of Jarlsberg on BMD and bone markers to OP patients.
* To compare daily intake of Ca and vitamin D with and without OED of Jarlsberg on Time-to-Osteoporotic (TTO) treatment is recommended.

Study population consists of OP-patients of post-menopausal women and men above 55 years of age. OP patients are defined as patients with a T-score below 0.0, but larger than -2.5.

Women in post-menopausal age have a daily OED Jarlsberg of 45 gram and men in the same age interval have a daily OED of 55 gram.

The cheese will be delivered in package of 250 gram with slices of 15.625gram. 45 gram represents 3 slices; 55 gram 4 slices. All the included patients will receive 20µg vitamin D and 1000 mg Ca. Half of the patients will receive vitamin D and Ca-tablets plus Jarlsberg cheese (Treatment group I) and other half only vitamin D and Ca-tablets (Treatment group II).

Design: The study will be performed as a randomized, single-blinded Norwegian multicentre trial with stratified semi-cross-over design with gender and site as stratification factors.

Patients included in the study will be allocated to one of the two treatment groups by block randomization with random block size between 2 and 6.

Main variables: The main response variable will be the change in Bone Mineral Density (BMD).The secondary variables will be total Osteocalcin (tOC), carboxylated osteocalcin (cOC), the osteocalcin ratio and different bone markers (BM). Additionally, the K2 vitamers MK-7, MK-8, MK-9, and MK-9(4H) will be used as explanatory variable together with the Interleukins IL-1β, IL6, IL8, IL10 and the Cytokines TNF-α, NF-ƙβ (RANK-L), OPG and TGF-β . Diet registration as controlling variables and HbA1C, Lipids, biochemical variables will be used as supporting variables. The Common Terminology Criteria for Adverse Events version 4.0 (CTCAE) will be used for registration of Adverse Events (AE) and toxicity score at every investigation visit.

Study procedure: Participants, who fulfil the inclusion criteria, do not meet any of the exclusion criteria and willing to give informed consent to participate will be included in a screening period of one week. During this screening week, all the possible participants will receive 40µg vitamin D and 500 mg Ca tablets per day, but asked not to eat Jarlsberg cheese.

BMD measurements will be taken at the start of the screening week. Patients with a negative BMD T-score >-2.5 will be included in the study. All demographic data, social factors, history of disease and vital signs will be recorded at baseline. The participating patients will be given a Diet-App on the web or mobile phone for registration of the daily food intake during four first consecutively days after baseline. Blood samples for measurements of Osteocalcin, BM and vitamin K will be taken fastening in the morning. Additionally, blood samples for measuring biochemical variables, HbA1C, Lipids, Interleukins and Cytokines, will be recorded. The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 used for measuring and classifying the tolerability and toxicity will be recorded as well. The patients will be given a compliance & activity form and asked to write down the daily intake of treatment medicine, Jarlsberg cheese and hours of physical activities.

Clinical part: The patients will be allocated (1:1) to vitamin D + Ca-tablets ± OED of Jarlsberg cheese. All the participants will get new delivery of vitamin D and Ca-tablets every four weeks. The patients allocated to Jarlsberg will additionally receive Jarlsberg cheese. The patients will receive a compliance & activity form and asked to fill in every day. All the patients meet for new visits at week4, week 16, and week 32. Patients allocated to only vitamin D + Ca tablets at baseline well additionally meet for visits at week 20 and week 48. At all these visits blood samples for measurement of Osteocalcin, BM and PTH will be drawn fasting in the morning, and concomitant medication and treatment compliance recorded.

The main visit will be performed every 16 weeks. New DXA screening will be performed. Patients obtaining a BMD T-score ≤ -2.5 will discontinue the study and switched to antiresorptive treatment plus daily OED of Jarlsberg cheese. The daily food intake during four consecutively days will be recorded on the Diet-App. Blood samples for measurements of Osteocalcin, CTX-1, PINP, BALB and PTH will be drawn fastening in the morning at every visits. Furthermore, blood samples for measuring and biochemical variables, HbA1C and Lipids, will be recorded. The CTCAE will be recorded as well.After the first 16 weeks, the patients allocated to only Ca + vitamin D will additionally receive OED of Jarlsberg cheese out the study. The visit at Week 32 and Week 48 will be the last observation for the patients initially allocated to Jarlsberg and controls, respectively. In addition to the mentioned variables, blood samples for measurement of Interleukins and Cytokines will be performed. All the patients completed the study will be offered to continue the daily intake of OED Jarlsberg cheese. These patients will be followed up one year after the last visit with a new DXA and a blood sampling for measurements of Osteocalcin level and BM.

Sample size:

With a significance level of 5%, a power of 90% and a Clinically Relevant Difference (CRD) of one time the Standard Deviation in change of BMD, at least 24 patients in each group must finalize the study. With an expected drop-out rate of 25%, 30 patients in each group must be included.

ELIGIBILITY:
Inclusion Criteria:

* Osteopeni patients (OP) of both genders above 55 years of age. OPs are defined as patients with T-score below 0.0 but larger than -2.5.

Exclusion Criteria:

* • Eating disorder

  * Known gastrointestinal disorder.
  * Abnormal liver or kidney function.
  * Diabetes mellitus type I.
  * Diabetes type II without sufficient control.
  * Suffering from verified cancer.
  * Under systemic treatment with corticosteroids or other immunosuppressive drugs the last 3 weeks before start of the trial treatment.
  * Under active antiresorptive treatment or anabolic treatment.
  * Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
  * Known milk product allergy.
  * Not able to understand information.
  * Do not want or not able to give written consent to participate in the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Post menopausal women
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | Week 0
  g/cm2
Bone Mineral Density | Week 16
  g/cm2
Bone Mineral Density | Week 32
  g/cm2
Bone Mineral Density | Week 48
  g/cm2

SECONDARY OUTCOMES:
Osteocalcin | week 0
  ng/ml
Osteocalcin | week 4
  ng/ml
Osteocalcin | week 16
  ng/ml
Osteocalcin | week 20
  ng/ml
Osteocalcin | week 32
  ng/ml
Osteocalcin | week 48
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 0
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 4
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 16
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 20
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 32
  ng/ml
Procollagen type 1 N-terminal propeptide (PINP) | Week 48
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 0
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 4
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 16
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 20
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 32
  ng/ml
Cross-linked C-telopeptide type I collagen (CTX) | week 48
  ng/ml
Bone specific ALP (BALB) | Week 0
  ng/ml
Bone specific ALP (BALB) | Week 4
  ng/ml
Bone specific ALP (BALB) | Week 16
  ng/ml
Bone specific ALP (BALB) | Week 20
  ng/ml
Bone specific ALP (BALB) | Week 32
  ng/ml
Bone specific ALP (BALB) | Week 48
  ng/ml

OTHER OUTCOMES:
Vitamin K2 | Week 0
  ng/ml
Vitamin K2 | Week 16
  ng/ml
Vitamin K2 | Week 32
  ng/ml
Vitamin K2 | Week 48
  ng/ml
Interleukin IL-1β, IL6, IL8, IL10 | Week 0
  ng/ml
Interleukin IL-1β, IL6, IL8, IL10 | Week 32
  ng/ml
Interleukin IL-1β, IL6, IL8, IL10 | Week 48
  ng/ml
Cytokine TNF-α, NF-ƙβ (RANK-L), OPG, TGF-β | Week 0
  ng/ml
Cytokine TNF-α, NF-ƙβ (RANK-L), OPG, TGF-β | Week 32
  ng/ml
Cytokine TNF-α, NF-ƙβ (RANK-L), OPG, TGF-β | Week 48
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Whist, PhD, Study Director — Tine
Locations (1):
- Meddoc, Skjetten, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT05787808/Prot_000.pdf